CLINICAL TRIAL: NCT00283816
Title: Metabolic Impact of Oral Contraceptives With or Without Metformin in Obese Adolescents With Polycystic Ovary Syndrome (PCOS)
Brief Title: Impact of Metformin in Teens With Polycystic Ovary Syndrome (PCOS) on Oral Contraceptive Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Kathleen M. Hoeger, MD, Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RSRB-00012501; GCRC#1083
Record Dates: First submitted 2006-01-27; First posted 2006-01-30 (Estimated); Results first posted 2011-07-13 (Estimated); Last update posted 2015-05-15 (Estimated); Status verified 2011-04

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Polycystic Ovary Syndrome; Overweight Adolescent Girls; Irregular Menstrual Cycles
MeSH Terms: conditions — Polycystic Ovary Syndrome; Menstruation Disturbances | interventions — Metformin; Contraceptives, Oral; Glucose Tolerance Test; Absorptiometry, Photon

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): metformin
  Interventions: Drug: Metformin; Drug: Oral Contraceptive Pill; Behavioral: Lifestyle Management Program; Behavioral: Quality of Life Questionnaire; Procedure: Oral Glucose Tolerance Test; Procedure: Blood work; Procedure: Abdominal Ultra Sound; Procedure: Dual-energy x-ray absorptiometry (DEXA scan)
- 0 (Placebo Comparator): placebo
  Interventions: Drug: Oral Contraceptive Pill; Behavioral: Lifestyle Management Program; Behavioral: Quality of Life Questionnaire; Procedure: Oral Glucose Tolerance Test; Procedure: Blood work; Procedure: Abdominal Ultra Sound; Procedure: Dual-energy x-ray absorptiometry (DEXA scan); Drug: placebo

INTERVENTIONS:
Drug: Metformin — Metformin 500 mg. tabs 2 tabs BID for duration of study
  Other Names: Metformin Hydrochloride Tablets, 500 mg.; manufacturer: Mylan Pharmaceuticals, Morgantown, WV
  Arms: 1
Drug: Oral Contraceptive Pill — Yasmin, drospirenone and ethinyl estradiol 28 tablets
  1 tab daily for duration of study
  Other Names: Yasmin 28 tablets; Manufacturer: Berlex, Montville, NJ 07045
Behavioral: Lifestyle Management Program — Subjects and a parent/guardian will participate in a series of classes for training in diet, exercise & behavior modification skills on a regular weekly basis over the 24 week study
Behavioral: Quality of Life Questionnaire — Quality of Life questionnaire designed for women with Polycystic Ovary Syndrome. Questions concern health and health related issues Performed twice during study, at baseline and conclusion
Procedure: Oral Glucose Tolerance Test — Insulin response to a glucose challenge in an oral glucose tolerance test (OGTT), as measured by area under the curve (AUC). In this study we will administer an OGTT and calculate the AUC as a measure of insulin resistance.
  Performed twice during study, at baseline and conclusion
Procedure: Blood work — Initial and conclusion blood draws include; comprehensive metabolic profile, CBC and platelet,hormonal assessment and lipids.
Procedure: Abdominal Ultra Sound — transabdominal transducer, which contains integrated software for volume calculation will be used to assess ovarian volume.
  Performed twice during study, at baseline and conclusion
Procedure: Dual-energy x-ray absorptiometry (DEXA scan) — Dual-energy x-ray absorptiometry (DEXA) will be used to assess percent body fat Performed twice during study, at baseline and conclusion
Drug: placebo — placebo capsules, two capsules BID
  Other Names: placebo formulation: 240 mg. lactose powder USP; in size 3 capsules from Capsugel
  Arms: 0

SUMMARY:
Oral contraceptives are known to improve menstrual cycles and symptoms in PCOS, however may increase cholesterol. Metformin, a drug to improve insulin resistance, may benefit metabolic state. This study is to determine whether metformin added to oral contraceptive therapy in adolescent women with PCOS improves metabolic state.The study will also test a lifestyle improvement program to reduce weight.

DETAILED DESCRIPTION:
Polycystic Ovary Syndrome (PCOS) is a heterogeneous condition characterized by chronic anovulation and androgen excess that occurs in 4-8% of unselected adult women. Although signs and symptoms of the disorder typically appear at the time of puberty, diagnosis is often delayed until adulthood. At least 50% of adult women with PCOS are obese, resulting in a more severe clinical picture. Obesity among adolescents has been increasing in recent years, with overrepresentation of females who show evidence of hyperandrogenism and irregular periods, suggesting an association of obesity and PCOS at an early age. Recent data, however, have drawn attention to the long-term risks of PCOS, including diabetes and cardiovascular disease. Insulin resistance plays a critical role in the pathophysiology of PCOS and is thought to be the metabolic abnormality most closely linked to an increased risk of diabetes and heart disease. Traditional treatments with oral contraceptives are associated with reduction in serum androgens and improvements in menstrual cycles in adolescents with PCOS, however these have not been well-studied in obese adolescents. Oral contraceptives may worsen the dyslipidemia seen in obese women with PCOS and do not address the insulin resistance. Metformin, an insulin sensitizing agent, has been shown to improve metabolic features of PCOS, but combination therapy with oral contraceptives has never been studied in the obese adolescent with PCOS.

The major hypothesis of this proposal is that metformin will improve the metabolic profile of obese adolescent girls with PCOS treated with oral contraceptives. Additionally, a secondary hypothesis will be that compliance with a concurrent lifestyle modification program with be associated with the most significant improvements.

ELIGIBILITY:
Inclusion Criteria:Age 12-18 years; Menstrual irregularity; Overweight; Must be able to swallow capsules; At lease 6 months since onset of first menstrual cycle.

Exclusion Criteria:Diabetes; Kidney or Liver disease; Tobacco use; Depression or Bipolar Disease; Contraindication to exercise; Weight > 300 lbs.

Ages: 12 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2006-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Hoeger, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Metformin: Subjects given 2000mg of metformin in addition to oral contraceptive and a lifestyle program
- Placebo: Subjects given a placebo in addition to oral contraceptive and lifestyle program
Period: Overall Study
Arm/Group | Metformin | Placebo
Started | 18 | 18
Completed | 16 | 16
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin | Placebo | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 18 | 18 | 36
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.7 (1.6) | 15.8 (1.6) | 15.1 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 36
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 18 | 36

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Abdominal Fat as Measured by Waist Circumference.
Description: Change in waist circumference measured in cms used as a measure of abdominal adiposity, pre minus post intervention
Time Frame: baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: cm
Groups:
- Metformin: 2000mg of metformin in addition to oral contraceptive
- Placebo: placebo pill in addition to oral contraceptive pill
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 16 | 16
cm | -3.9 (8.6) | -1.4 (10.9)

2. Secondary Outcome: Change in Weight Post Minus Pre Intervention.
Description: Body mass index change in adolescents enrolled in lifestyle intervention program
Time Frame: baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: kg/m^2
Groups:
- Metformin: metformin 2000mg in addition to oral contraceptive
- Placebo: placebo pill in addition to oral contraceptive
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 16 | 16
kg/m^2 | -1.9 (4.7) | -1.2 (4.5)

3. Secondary Outcome: Total Testosterone Change
Description: Change in total testosterone post minus pre intervention
Time Frame: baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 16 | 16
ng/dL | -57.7 (21.7) | -27.6 (30.1)

4. Secondary Outcome: Change in Sex Hormone Binding Globulin (SHBG)
Description: SHBG concentration post minus pre-intervention
Time Frame: baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 16 | 16
nmol/L | -73.4 (31.9) | -58 (34.3)

ADVERSE EVENTS:
Arm/Group | Metformin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No